CLINICAL TRIAL: NCT01412346
Title: Health Effects of a Nordic Diet Rich in Plant-based Foods and Fish
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Finnish Institute for Health and Welfare (Other Government)
Collaborators: Academy of Finland (Other); University of Oslo (Other)
Responsible Party: Principal Investigator, Iris Erlund, PhD., senior researcher, Finnish Institute for Health and Welfare
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NPHIKTL_022011
Record Dates: First submitted 2011-08-03; First posted 2011-08-09 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Prehypertension; Hypertension
Keywords: human; clinical trial; dietary intervention study; blood pressure; cardiovascular biomarkers; nutritional biomarkers; gene expression
MeSH Terms: conditions — Prehypertension; Hypertension | interventions — In Situ Hybridization, Fluorescence

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Plant-based food and fish with salt restr. (Active Comparator): The subjects consume plant based foods (fruits, berries, vegetables, whole grain) and fish in addition to a salt-restricted diet. Intake of salt is normal to high for 8 weeks and low for 8 weeks (subjects receive salt and placebo capsules in a crossover design).
  Interventions: Other: Effects of a Nordic diet rich in plant-based foods and fish
- Diet with salt restriction (Placebo Comparator): The subjects follow a salt-restricted diet. Intake of salt is normal to high for 8 weeks and low for 8 weeks (subjects receive salt and placebo capsules in a crossover design).
  Interventions: Other: Effects of a Nordic diet rich in plant-based foods and fish

INTERVENTIONS:
Other: Effects of a Nordic diet rich in plant-based foods and fish — The intervention lasts for 20 weeks and it includes dietary counseling concerning salt restriction. Key foods are provided to the subjects.

SUMMARY:
The purpose of this study is to investigate the effects of a Nordic diet rich in plant-based foods and fish on indicators of cardiovascular disease risk at two different levels of salt intake.

The study is a 20-wk randomized controlled crossover trial. The subjects follow a salt-restricted diet during the study. The study begins with a 4-wk run-in phase for all subjects. After that the subjects are randomly allocated to one of two groups. Group 1 consumes a healthy Nordic low-salt diet enriched with plant-based foods and fish for 16 weeks. Group 2 consumes a low-salt diet for 16 weeks. During the 16 weeks, both groups receive salt and placebo capsules in a double-blind, crossover fashion (8+8 weeks).

ELIGIBILITY:
Inclusion Criteria:

* prehypertension or hypertension (systolic blood pressure 130-159 mmHg or diastolic blood pressure 85-99 mmHg)

Exclusion Criteria:

* smoking
* regular use of medications
* intestinal disorders
* symptomatic cardiovascular disease
* obesity (BMI>35 kg/m2)
* vegetarianism
* high intake of alcohol
* allergy to fish
* pregnancy

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2011-01; Primary Completion 2012-06 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in systolic and diastolic blood pressure after treatments | 12 and 20 weeks

SECONDARY OUTCOMES:
Change from baseline in PFA-100 measurements after treatments | 12 and 20 weeks
Change from baseline in biomarkers of cardiovascular disease risk after treatments | 12 and 20 weeks
Change from baseline in nutritional biomarkers after treatments | 12 and 20 weeks
Change from baseline in blood cell gene expression after treatments | 12 and 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Iris Erlund, Dr., Study Director — Finnish Institute for Health and Welfare; Antti Jula, Dr., Study Director — Finnish Institute for Health and Welfare
Locations (1):
- National Institute for Health and Welfare, Helsinki, Finland

REFERENCES:
- [Derived] Niiranen T, Erlund I, Jalkanen S, Jula A, Salmi M. Effects of altered salt intake and diet on cytokines in humans: A 20-week randomized cross-over intervention study. Eur J Immunol. 2023 Jan;53(1):e2250074. doi: 10.1002/eji.202250074. Epub 2022 Nov 20. PMID 36330564